CLINICAL TRIAL: NCT00954226
Title: Phase Ib Study of Erlotinib Prior to Surgery in Patients With Head and Neck Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2008-0137; NCI-2012-01639 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); NCI-2010-01142; 2008-0137 (Other: M D Anderson Cancer Center)
Record Dates: First submitted 2009-08-06; First posted 2009-08-07 (Estimated); Last update posted 2025-09-05 (Actual); Status verified 2025-08

CONDITIONS: Recurrent Head and Neck Carcinoma; Recurrent Salivary Gland Carcinoma; Recurrent Skin Carcinoma; Skin Squamous Cell Carcinoma
MeSH Terms: conditions — Salivary Gland Neoplasms | interventions — Erlotinib Hydrochloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm I (standard-dose erlotinib hydrochloride) (Experimental): Patients receive standard-dose erlotinib hydrochloride PO QD for 2-3 weeks (up to 8 weeks if surgery is delayed).
  Interventions: Drug: Erlotinib Hydrochloride; Other: Laboratory Biomarker Analysis
- Arm II (high-dose erlotinib hydrochloride) (Experimental): Patients receive high-dose erlotinib hydrochloride PO QD for 2-3 weeks (2-8 weeks for current smokers or up to 8 weeks if surgery is delayed).
  Interventions: Drug: Erlotinib Hydrochloride; Other: Laboratory Biomarker Analysis

INTERVENTIONS:
Drug: Erlotinib Hydrochloride — Given PO
  Other Names: Cp-358,774; OSI-774; Tarceva
Other: Laboratory Biomarker Analysis — Correlative studies

SUMMARY:
This randomized phase Ib trial studies standard-dose or high-dose erlotinib hydrochloride before surgery in treating patients with head and neck cancer. Erlotinib hydrochloride may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the effects of erlotinib (erlotinib hydrochloride) 150 mg/day (standard dose) and 200 mg/day or 300 mg/day (high-dose) on the phosphorylation of AKT protein downstream from epidermal growth factor receptor (EGFR).

SECONDARY OBJECTIVES:

I. To assess the safety and tolerability of erlotinib 150 mg/day (standard dose) and 200 mg/day or 300 mg/day (high-dose).

II. To correlate the effects of erlotinib on the phosphorylation of AKT with the immunohistochemical expression level of EGFR and the level of amplification of the EGFR gene as determined by fluorescent in situ hybridization (FISH).

III. To evaluate the preliminary response rate with a short course of erlotinib.

IV. To evaluate changes in the activation status of proteins downstream from EGFR and other receptor tyrosine kinases and in markers of epithelial to mesenchymal transition.

V. To evaluate changes in blood-based biomarkers. VI. To evaluate the effects of a higher dose of erlotinib (300 mg/day) in current smokers.

TERTIARY OBJECTIVES:

I. To evaluate EGFR gene copy number by fluorescent in situ hybridization. II. To evaluate immunohistochemistry, western blotting and reverse phase protein lysate arrays to assess the activation (usually phosphorylation) status of other downstream proteins from EGFR and other receptor tyrosine kinases (these will include, but are not restricted to: EGFR itself, phosphatidylinositol 3 Kinase [PI3K], AKT, mammalian target of rapamycin [mTOR], glycogen synthase kinase 3 [GSK3], p70 ribosomal S6 kinase [p70S6K], S6, 4E-binding protein 1[4E-BP1], MEK1/2, mitogen-activated protein kinase [MAPK], p38, -c-Jun N-terminal kinase [JNK], insulin-like growth factor 1 receptor [IGF-1R], IGF-2R, mesenchymal epithelial transition [MET], hypoxia-inducible factor [HIF]) both before and after treatment with erlotinib.

III. To evaluate immunohistochemical expression levels of markers of epithelial to mesenchymal transition (these will include, but are not restricted to: e-cadherin and vimentin).

IV. To study blood-based biomarkers of interest, which will include (but are not restricted to): trough levels of erlotinib and its metabolites, a panel of 59 cytokine and angiogenic factors measured by available Luminex multiplex beads kits (Bio-Plex 27-Plex & 23-Plex Kits [Bio-Rad, Hercules, CA] and Human cardiovascular disease [CVD] Biomarker Panel 1 kit [Linco Research, Inc., St, Charles, MO]) as well as validated enzyme-linked immunosorbent assays for soluble vascular endothelial growth factor receptor 1(VEGFR1), VEGFR2 (Invitrogen, Carlsbad, CA), total IGF-1, IGF-2, insulin-like growth factor-binding protein (IGFBP3) (DSL, Webster, TX), and osteopontin (R&D Systems, Minneapolis, MN).

V. To evaluate whole genome sequencing and/or sequencing of specific genes of interest, analysis of gene copy number, messenger ribonucleic acid (mRNA) expression profiles, non-coding RNA expression profiles, single nucleotide polymorphisms, deoxyribonucleic acid (DNA) methylation profiles, immunohistochemistry of proteins of interest to head and neck cancer biology, and proteomics in tumor tissue and/or normal tissue (including blood) before and after treatment with erlotinib.

OUTLINE: Patients are randomized to 1 of 2 treatment arms.

ARM I: Patients receive standard-dose erlotinib hydrochloride orally (PO) once daily (QD) for 2-3 weeks (up to 8 weeks if surgery is delayed).

ARM II: Patients receive high-dose erlotinib hydrochloride PO QD for 2-3 weeks (2-8 weeks for current smokers or up to 8 weeks if surgery is delayed).

After completion of study treatment, patients are followed up within 30 days.

ELIGIBILITY:
Inclusion Criteria:

* Patients with histologically confirmed cancer of the head and neck. Patients with salivary gland tumors and squamous cell carcinomas of the skin are also eligible. (Note: Any patient with a diagnosis of aggressive squamous cell carcinoma of the skin and determined to be surgically resectable will be considered for eligibility. These patients are typically seen in the Head & Neck surgery clinic and decisions for study consideration will be based on consultations with the department of Head & Neck surgery.)
* The patient must have biopsy-accessible disease.
* Patients must be surgical candidates (either definitive or palliative setting).
* Patients may have received prior therapy including cytotoxic chemotherapy (e.g. platinum drugs and taxanes) and radiation therapy.
* Patients must have a performance score (ECOG) of 0-2.
* Patients should have adequate bone marrow function, as defined by peripheral granulocyte count of >/= 1,000/mm³, and a platelet count of >/= 50,000/mm³.Patients must have adequate liver function with a bilirubin </= 1.5 times the upper limit of normal (ULN). Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) must be </= 2 x the ULN and alkaline phosphatase must be </= 2 x ULN.
* Patients should have adequate renal function (serum creatinine </= 1.5 x ULN).
* Age >/= 18 years
* Ability to understand and the willingness to sign a written informed consent document indicating that they are aware of the investigational nature of the study, in keeping with institutional policy
* Women of childbearing potential must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation. Childbearing potential will be defined as women who have had menses within the past 12 months,who have not had tubal ligation or bilateral oophorectomy. Should a woman become pregnant or suspect that she is pregnant while participating in this study,she should inform her treating physician immediately.The patient,if a man,agrees to use effective contraception or abstinence.

Exclusion Criteria:

* Patients with prior exposure to small molecule tyrosine kinase inhibitors or EGFR-targeted antibodies within the past 6 months.
* Patients for whom, in the opinion of the treating surgeon, the administration of erlotinib would cause a deleterious delay in surgical treatment.
* Patients with uncompensated congestive cardiac failure.
* Patients with an organ allograft.
* Patients with a serious concurrent infection or illness including, but not limited to, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness that could limit compliance with study requirements.
* Female patients who are pregnant or breastfeeding
* Patients currently on chemotherapy, immunotherapy, or therapy with monoclonal antibodies or other investigational agents with anti-tumor activity

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2009-08-05 (Actual); Primary Completion 2025-04-30 (Actual); Study Completion 2025-04-30 (Actual)

PRIMARY OUTCOMES:
Change in modulation of the biomarker phospho-Akt in tumor specimens | From baseline to surgery
  Modulation of phospho-Akt (difference in immunohistochemistry [IHC] score between the surgical specimen and the baseline biopsy) will be compared between the two treatment arms (i.e., standard-dose and high-dose) with the use of Wilcoxon rank sum test.

CONTACTS AND LOCATIONS:
Overall Officials: Xiuning Le, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: M D Anderson Cancer Center — http://www.mdanderson.org

DOCUMENTS (1):
  • Informed Consent Form (2018-04-02): https://cdn.clinicaltrials.gov/large-docs/26/NCT00954226/ICF_000.pdf